CLINICAL TRIAL: NCT01617278
Title: A Randomized Controlled Trial Comparing High-definition White Light Colonoscopy to I-Scan Enhanced Colonoscopy for Adenoma Detection in a Population at Increased Risk of Colorectal Cancer. (A Pilot Study)
Brief Title: I-Scan Versus High-definition White Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Robert Hilsden, Associate Professor, Department of Medicine & Research Director, Colon Cancer screening Centre, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23474-P
Record Dates: First submitted 2012-06-04; First posted 2012-06-12 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer
Keywords: Colonoscopy; I Scan; High definition white light; Adenomas
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- I-Scan 1 (Experimental): I-Scan 1 modality will be used by the endoscopist for the entire procedure
  Interventions: Device: I-Scan 1
- HD Colon (Experimental): High definition white light modality will be used by the endoscopist for the entire procedure
  Interventions: Device: HD Colon
- I-scan 2 (Experimental): I-Scan 2 modality will be used by th endoscopist through out the procedure
  Interventions: Device: I-Scan 2

INTERVENTIONS:
Device: I-Scan 1 — I-Scan 1 has contrast enhancement (CE)and surface enhancement (SE). SE mode highlights light-dark contrast thereby providing more mucosal surface detail.CE mode digitally adds blue to darker areas providing detailed imaging of subtle mucosal irregularities.
  Arms: I-Scan 1
Device: HD Colon — High definition white light
  Arms: HD Colon
Device: I-Scan 2 — I-Scan 2 has contrast enhancement (CE), surface enhancement (SE) and tone enhancement (TE). SE mode highlights light-dark contrast thereby providing more mucosal surface detail.CE mode digitally adds blue to darker areas providing detailed imaging of subtle mucosal irregularities.TE provides a uniform colour image and is intended for detailed inspection of distinct lesions.
  Arms: I-scan 2

SUMMARY:
The purpose of the study is to assess whether the use of I-scan during colonoscopy leads to an increased yield of adenomas in the colon among a population at increased risk for CRC.

Primary Outcome:

To estimate the mean number of adenomas per colonoscopy for both high definition white light colonoscopy and I-scan enhanced colonoscopy

Secondary Outcomes:

1. To estimate the recruitment rate
2. Number of adenomas detected in the right colon during the second look

DETAILED DESCRIPTION:
Colorectal Cancer is the third most common cause of cancer in Canada with an estimated lifetime risk of developing the disease of 6-7%. Each year there are approximately 21,000 new cases and 9,100 deaths attributable to this disease. Colonoscopy is one of several methods recommended for CRC screening by current guidelines. While colonoscopy is the most invasive, it offers high diagnostic accuracy and ability for therapy (biopsy and removal of adenomas) compared to other modalities. The emerging evidence regarding missed neoplastic lesions with colonoscopy has resulted in quality initiatives designed to improve colonoscopy performance. I-Scan (Pentax, Montvale, NJ) is a new method that uses post processing computer algorithms to revise the standard white light to highlight pit patterns and vascular surface patterns.The relevant I-scan settings in the colon are I-scan 1 and I-scan 2. The primary objective of the study is to compare the adenoma detection rate in the right colon using High-definition white light colonoscopy versus I-scan enhanced colonoscopy.

All patients referred for a screening colonoscopy at Forzani and MacPhail Colon Cancer Centre will be considered for enrollment.All eligible patients that are not part of another research study will be approached for enrollment into the study. During the pre-assessment at the clinic a study assistant will contact all the eligible patients to describe the study and provide an "Invitation to participate in a Research study" form. The study assistant will obtain a final consent if they agree. Those not interested will simply receive the Centre's standard protocol. There will be no coercion of any sort. Following Informed Consent, treatment allocation through computer generated randomization will be revealed. Patients will be allocated to one of the three study arms (HD Colon, I-scan 1 and I-Scan 2). Patients will receive a standard bowel preparation: Split dose Polyethylene Glycol (PEG) (2L at noon + 2L at 8 PM the day before) for morning procedures or (2L at 8Pm the day before and 2L at five hours before the procedure on the day of colonoscopy) for afternoon procedure. certified gastroenterologists will perform all of the procedures with the assistance of a nurse. The planned "second look" of the right colon will involve withdrawing from the Cecum to Hepatic flexure, then re-inserting to Cecum and finally withdrawing through the entire colon. The physician performing the procedure will then fill a "Colonoscopy Report Form" including the number of polyps detected, size, shape, polypectomy method and cleanliness of the bowel.

ELIGIBILITY:
Inclusion Criteria:

* All increased risk patients (Patients with family history or personal history of Colon Polyps or Colon Cancer and FOBT positive) referred for a screening colonoscopy at the Forzani and MacPhail Colon Cancer Centre will be considered for enrollment

Exclusion Criteria:

* Average risk patients
* Previous Colon surgery
* Hereditary Polyposis syndromes
* Suspected polyps or CRC before colonoscopy that have been suggested by another modality (Barium enema, Virtual colonoscopy, Flexible Sigmoidoscopy)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Mean number of adenomas per colonoscopy | Colonoscopy report form provided to the physician will be filled out and collected after the procedure (1 hour). All polyps reviewed by pathologist (1 week).
  The "Colonoscopy Report Form" completed by the Physician helps to assess the number of polyps and a endoscopic description (location, size, shape) of these lesions including. Following formal review by the pathologist the polyp classification (e.g. whether it is an adenoma) is determined.

SECONDARY OUTCOMES:
Number of adenomas detected in the right colon during the second look | Second look in the right colon and finally withdrawing through the entire colon (approximately 5 min)
  The planned "Second Look" of the right colon will involve withdrawing from the cecum to hepatic flexure, then re-inserting to the cecum and finally withdrawing through the entire colon. This is to determine if a "Second Look" in the right colon increases the mean number of adenomas detected compared with a single inspection irrespective of the imaging modality.
To estimate the recruitment rate | Upto 8 months
  Recruitment rates will be reported as follows:
  1. No. of patients given the study invitation letter
  2. No. of patients who return the form as interested
  3. No. of patients who provided informed consent
  4. No. of patients who complete the study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hilsden, MD, Principal Investigator — Faculty of Medicine, University of Calgary
Locations (1):
- Forzani & MacPhail Colon Cancer Screening Centre, Alberta Health Services, Calgary, Alberta, Canada